CLINICAL TRIAL: NCT00178555
Title: A Comparison of Laryngoscopy Techniques Using the Video Laryngoscope and the Traditional Macintosh Laryngoscope in Patients Who May be Difficult to Intubate
Brief Title: Comparison of the Video and Macintosh Laryngoscope in Patients Who May be Difficult to Intubate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Principal Investigator, Carin A. Hagberg, Professor and Chairman, Joseph C. Gable, M.D., Endowed Chair, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HSC-MS-03-082
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Intubation, Endotracheal
Keywords: Endotracheal Intubation, Video Laryngoscopy

INTERVENTIONS:
Device: DCI Video Intubation System-Macintosh Laryngoscope
Device: Macintosh Laryngoscope

SUMMARY:
The purpose of this study is to determine if the Video Laryngoscope (VL) is a useful instrument in patients at risk for difficult intubation. We will compare this device to the traditional Macintosh Laryngoscope.

DETAILED DESCRIPTION:
Despite improvements made to the traditional laryngoscope blade since its invention, occasionally intubation of the trachea cannot be accomplished with facility, even in patients with anatomy that does not predict difficult intubation. It is estimated that endotracheal intubation is performed on some 8 million patients per year in the United States. Of these endotracheal intubations, approximately 80% are performed by direct laryngoscopy with transoral placement of the endotracheal tube (ET) into the trachea. There is fairly uniform reporting of the incidence of failed intubation in the literature; it occurs in approximately 0.05% or 1:2230 of surgical patients and in approximately 0.13% to 0.35%, or 1:750 to 1:280, of the obstetric patients. The incidence of unsuspected difficult intubation is estimated to be higher at 3%. One factor that contributes to difficult intubation is poor visualization.

The VL is designed to optimize visualization by presenting to the operator an enlarged video image of airway structures. In contrast, using conventional laryngoscopy, anesthesiologists have only a "keyhole" view of the airway structures; a view that may be further obscured during attempts to pass the ET.

The VL consists of a laryngoscope handle and Macintosh blade that have been modified to provide a video image of airway structures on a screen, which can be conveniently located directly in front of the anesthesiologist. A micro video module is contained in the modified handle. An image/light bundle is introduced into the standard blade. This system has been previously tested in which the consensus was that the device is extremely easy to learn to use because most anesthesiologists are familiar with the use of the Macintosh blade. It has also been useful in the instruction of laryngoscopy by non-anesthesiologists.

There are several potential advantages of a video image in the context of direct laryngoscopy. The system provides high quality video images that are enlarged on the video monitor for easier visualization. If laryngeal manipulation is required to improve visualization of laryngeal structures, the intubator and the person assisting can coordinate movements as they observe, simultaneously, the image on the video monitor. With the video image projected from the distal end of the laryngoscope blade, laryngeal structures are kept in view as the ET is passed through the oropharynx into the trachea.

Comparison: Video Laryngoscope as a conduit for possible difficult intubation compared to the traditional Macintosh blade.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* ASA I-III
* Presenting for elective surgery
* Requires general anesthesia
* Present as a possible difficult intubation (one or more of the following)

  1. history of difficult intubations
  2. morbid obesity
  3. small mouth opening (<3 fingerbreadths)
  4. limited neck mobility
  5. Mallampati classes II-III
  6. short thyromental distance (<6 cm)

Exclusion Criteria:

* Determined to be easily intubated (none of the factors listed above)
* Considered so difficult (i.e. Mallampati IV) that an awake intubation should be performed
* ASA IV and V

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
5 scale score of glottic view; Time and number of attempts required; Level of difficulty; Degree of irritation of the pharynx, epiglottis, and aryteniods

SECONDARY OUTCOMES:
Vital signs, oxygen saturation, and end-tidal carbon dioxide

CONTACTS AND LOCATIONS:
Overall Officials: Carin A. Hagberg, M.D., Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States